CLINICAL TRIAL: NCT03139955
Title: A Single Group, Non-randomised, Feasibility Study Investigating the Use of Bodytrak® for Post Elective Surgery Patient Monitoring in the High Dependency Unit
Brief Title: Bodytrak® Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Inova Design Solutions Ltd (Industry)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other); Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: BT01
Record Dates: First submitted 2017-04-21; First posted 2017-05-04 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Monitoring, Physiologic; Vital Signs; Sepsis; Altered Level of Consciousness
Keywords: Feasibility Study; Pre/Post-Operative Patient Monitoring; Continuous Patient Monitoring; Patient Deterioration Identification; Bodytrak; National Early Warning System; Patient Safety
MeSH Terms: conditions — Sepsis; Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bodytrak: This is a single group study. 8 participants will be recruited and will receive the same intervention of physiological data collection using Bodytrak.
  Interventions: Device: Bodytrak

INTERVENTIONS:
Device: Bodytrak — Bodytrak is a wireless earpiece which can monitor the user's vital signs such as tympanic (ear) temperature and heart rate. The earpiece is non-invasive and should fit comfortably within the right ear, similar to an earphone with an over-the-ear hook. Bodytrak is currently in a prototype stage. For further information please visit http://www.bodytrak.co

SUMMARY:
Bodytrak® is a wireless earpiece which can monitor the user's vital signs such as tympanic (ear) temperature and heart rate. The earpiece is non-invasive and should fit comfortably within the right ear, similar to an earphone with an over-the-ear hook. Bodytrak is currently in a prototype stage.

The purpose of this study is to assess the feasibility of conducting a trial investigating the integration of Bodytrak in an NHS (National Health Service) environment at Chelsea and Westminster Hospital; to collect patient vital sign data for the development of Bodytrak algorithms to detect the transition point of recovery/deterioration of health, as well as the level of consciousness; and to obtain nurse and patient feedback regarding their user experience of Bodytrak.

DETAILED DESCRIPTION:
BACKGROUND Sepsis claims many lives annually, and poses a substantial drain on NHS (National Health System) resources. The use of a 'track-and-trigger' monitoring system, or the National Early Warning System (NEWS) has reduced mortality rates in recent years, by detecting the early onset of Sepsis. However, the acquisition of vital signs, required as part of NEWS, is a manual, error-prone, and time consuming process. Therefore, scope exists for improvement in the care pathway by automation and subsequent improvements in reliability, staff productivity, and patient treatment outcomes.

Post-operative patients are typically monitored for a period of time before they are discharged. Potentially, patient safety can be further improved, and earlier discharge can be enabled by means of a continuous vital signs monitoring device, with algorithms that can track deterioration/recovery rate. This complementary information, together with the NEWS score, can then provide objective metrics to aid the attending physician. The primary objectives of this study are to assess the effectiveness of Bodytrak in monitoring patient health.

In addition, within the set of vital signs monitored by NEWS, it is most difficult to automate the measurement of the Level of Consciousness/Alertness (LOC). Therefore, one objective of the proposed project is to investigate the feasibility of developing an unobtrusive method for automatically measuring LOC, of patients who are not under the influence of general anesthesia, which leads to the introduction of Bodytrak. Bodytrak® is a non-invasive, wireless ear-based device which can continuously monitor physiological parameters including tympanic temperature, photoplethysmography (PPG) derived heart rate and heart rate variability and accelerometer based motion metrics. The earpiece should fit comfortably within the right ear, similar to a earphone.

To this end, the physiological and biomechanical signals required for LOC algorithm development will be acquired using Bodytrak®. Automating the measurements of two other vital signs - Tympanic temperature and heart rate, will be carried out using Bodytrak® as well. Since these vitals are important predictors of Sepsis, and because they are currently part of the NEWS framework, providing reliable means of measurement, and automating the acquisition process is consistent with the goal of improving patient safety and staff productivity. As an important part of the study, these primary vital signs will be evaluated against validated medical devices.

Further, critical to eventual improvement of the care pathway by means of Bodytrak® is the feedback that can be gathered from both patients and clinical staff, since they are the end users of the system. If this application is approved, Inova intends to work closely with its partner, Chelsea and Westminster Hospital, in order to gather information necessary for the integration of Bodytrak® into the NEWS framework.

TRIAL DESIGN The trial is a non-blind, non-randomised single group feasibility study. 8 participants will be recruited who have scheduled elective surgery and aftercare in the HDU (high dependency unit). Patient participation will include 2 visits: a screening visit during a pre-clinic visit; and an intervention visit which will last approximately 2.5 days during their elective surgery in-patient stay in the high dependency unit. During their in-patient stay, participants will wear a Bodytrak earpiece during the day (for approximately 8 hours per day during the working hours of the research nurse), alongside continuous vital sign monitoring from hospital standard equipment (Philips Intellivue MP50 Monitor). The research nurse will carry out hourly checks on the patient to ensure the earpiece is not causing any discomfort. Patients will be asked to complete a feedback questionnaire regarding their experience of wearing Bodytrak. Research nurse's will also complete a feedback questionnaire regarding their use of Bodytrak.

While the sample size is admittedly small, note that the purpose of this study is NOT to validate Bodytrak® as a medical device, but rather to determine if it is feasible to devise reliable algorithms for reliably detecting the LOC and patient status, as well as to carry out a preliminary evaluation of the vital signs derived from Bodytrak®. A power analysis test will be carried out after the data collection has completed, in order to ascertain the validity of the statistical tests used and to determine if the sample size is sufficiently large. This would provide useful information for further studies that need to be carried out.

ELIGIBILITY:
Inclusion Criteria

In order to be able to participate in this study, an individual must meet all of the following criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female.
4. Age of ≥ 18 years at screening.
5. BMI between ≥19.0 and ≤30.0, inclusive.
6. An in-patient hospital stay in the high dependency unit of at least 2 days following elective general surgery at Chelsea and Westminster Hospital.
7. American Society of Anaesthesiologist (ASA) Physical status classification System 1-2
8. Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

1. Presence of a cardiac pacemaker.
2. Current or history of clinically significant cardiovascular disease, condition or abnormality including coronary artery disease, myocardial infarction, abnormal heart rhythms or arrhythmias, heart failure, heart valve disease, congenital heart disease, cardiomyopathy as determined by the physical exam or medical history review.
3. Use of the following cardiac drugs: beta blockers, calcium channel blockers, angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers/inhibitors or digitalis preparations within 3 months of Screening.
4. Current infection or condition of the right ear as determined by the Right Ear Exam or documented in medical history questionnaire, which may be exacerbated by the use of Bodytrak in the opinion of the investigator.
5. Patients who are on the ventilator and are persistently unconscious throughout their stay in the HDU.
6. Hypersensitivity or allergy to any of the Bodytrak materials that are in contact with the skin - SLA, PLA (3D printer resins), black Pro Flex 50 (Rubber), clear vacuum cast 40/55 shore silicone, and black anodised aluminium.
7. Patient known to have resistant organisms including Vancomycin-Resistant Enterococcus (VRE), Extended-Spectrum Beta-Lactamase (ESBL) & Methicillin-Resistant Staphylococcus aureus (MRSA), meaning Bodytrak would be unable to be cleaned using the approved cleaning protocol.
8. Any hearing impediment that, in the opinion of the investigator, would not be compatible with the use of Bodytrak.
9. Bodytrak not compatible to fit securely and correctly in the patient's right ear.
10. Participant unwilling to wear Bodytrak for the durations stated in the study protocol due to comfort and/or preference issues.
11. Pain reported during Right Ear Pain Assessment at screening
12. Currently participating in another clinical trial with an investigational or non-investigational drug or device, or has participated in another clinical trial within 3 months preceding Day 1.
13. Any condition that, in the opinion of the investigator, compromises the participant's ability to meet protocol requirements or to complete the study.
14. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
15. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre and post operative in-patients undergoing minor surgery and admitted for aftercare in the high dependency unit.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Bodytrak tympanic temperature data compared to gold standard hospital monitoring equipment | 2.5 days
  Establish if there are in-situ statistical and clinical significant differences between Bodytrak tympanic temperature and gold reference equipment used as part of standard care (tympanic thermometer). The extent of these differences will be measured using statistical tools such as 95% prediction interval, Bland-Altman plots, and correlation coefficients.
Accuracy of Bodytrak heart rate data compared to gold standard hospital monitoring equipment | 2.5 days
  Establish if there are in-situ statistical and clinical significant differences between Bodytrak heart rate and gold reference equipment used as part of standard care (3-lead ECG). The extent of these differences will be measured using statistical tools such as 95% prediction interval, Bland-Altman plots, and correlation coefficients.

SECONDARY OUTCOMES:
Level of alertness/consciousness (LOC) algorithm. | 2.5 days
  The efficacy of the LOC algorithm, as compared to the RASS consciousness scale will be measured using positive predictivity, sensitivity, and classification accuracy.

OTHER OUTCOMES:
Feedback from use of Bodytrak® in post-operative setting | Final study day (day 2.5)
  Questionnaires will be filled out by clinical staff operating the device, and patients who will be wearing it, in order to assess the usability of the device and find out desired features in the clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Vizcaychipi, Dr, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghasemi A, Zahediasl S. Normality tests for statistical analysis: a guide for non-statisticians. Int J Endocrinol Metab. 2012 Spring;10(2):486-9. doi: 10.5812/ijem.3505. Epub 2012 Apr 20. PMID 23843808
- [Background] Lin LI. A concordance correlation coefficient to evaluate reproducibility. Biometrics. 1989 Mar;45(1):255-68. PMID 2720055
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Gregoski MJ, Mueller M, Vertegel A, Shaporev A, Jackson BB, Frenzel RM, Sprehn SM, Treiber FA. Development and validation of a smartphone heart rate acquisition application for health promotion and wellness telehealth applications. Int J Telemed Appl. 2012;2012:696324. doi: 10.1155/2012/696324. Epub 2012 Jan 5. PMID 22272197
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] McNarry AF, Goldhill DR. Simple bedside assessment of level of consciousness: comparison of two simple assessment scales with the Glasgow Coma scale. Anaesthesia. 2004 Jan;59(1):34-7. doi: 10.1111/j.1365-2044.2004.03526.x. PMID 14687096
- See also: Further information regarding Bodytrak — http://www.bodytrak.co
- See also: J. Morrison, "Accessed 24 March 2017, Minimizing Bias in Experimental Design and Execution — https://neuronline.sfn.org/Articles/Professional-Development/2016/Minimizing-Bias-in-Experimental-Design-and-Execution